CLINICAL TRIAL: NCT07126327
Title: An Explorative Clinical Investigation to Understand the Clinical Benefits of Peristeen Light
Brief Title: Peristeen Light Explorative Clinical Investigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP378
Record Dates: First submitted 2025-06-27; First posted 2025-08-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Faecal Incontinence; Constipation - Functional
Keywords: trans anal irrigation
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploratory single-arm interventional investigation (Experimental): Prescription of Peristeen Light transanal irrigation system at enrolment to use for a 12 week test period
  Interventions: Device: Peristeen Light - trans anal irrigation system

INTERVENTIONS:
Device: Peristeen Light - trans anal irrigation system — Subjects naive to TAI will use Peristeen Light trans anal irrigation

SUMMARY:
The goal of this exploratory clinical investigation is to understand the clinical benefits of Peristeen Light in adult patients with faecal incontinence, chronic constipation and/or time-consuming bowel management procedures.

The primary objective is to evaluate changes in bowel-function when using Peristeen Light. Participants will use Peristeen Light for 12 weeks test period.

DETAILED DESCRIPTION:
The goal of this exploratory clinical investigation is to understand the clinical benefits of Peristeen Light in adult patients with faecal incontinence, chronic constipation and/or time-consuming bowel management procedures.

The primary endpoint is bowel function measured on a 10 cm Visual Analog Scale (VAS) at Baseline Visit and end of Clinical Investigation visit.

Participants will use Peristeen Light for 12 weeks test period.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent
* Is at least 18 years old
* Has full legal capacity
* Is able (assessed by investigator) and willing to adhere to clinical investigational procedures during clinical investigation-al duration
* Has access to and is able to use a smartphone
* Has constipation and/or faecal incontinence based on one or more of the following symptoms during the last 3 month: Straining in more than 25% of defecations, lumpy stools (Bristol Stool Type 1 and 2) in more than 25% of defecations, sensation of incomplete evacuation in more than 25% of defecations, sensation of anorectal obstruction/blockage in more than 25% of defecations, need to use manual maneuvers to facilitate defecation in more than 25% of defecations, fewer than three spontaneous bowel movements per week, loose stools are rarely present without use of laxatives, recurrent uncontrolled passage of faecal material (other words to describe this could be: Soiling, leak-age, passive faecal incontinence of flatus, mucus and/or stool)
* Is assessed (by investigator) to have a need for low-volume TAI minimum every other day

Exclusion Criteria:

* Is participating in any other clinical investigation during this investigation
* Has previously completed this investigation
* Is former or current user of transanal irrigation (low- and high volume)
* Has known hypersensitivity towards the device used in the investigation
* Is pregnant
* Has known anal stenosis
* Has active/recurrent colorectal cancer
* Has had anastomotic colorectal surgery within the last 3 months
* Has ischaemic colitis
* Has active inflammatory bowel disease
* Has acute diverticulitis or diverticular abscess
* Has medicine induced constipation (e.g. due to opioids)
* Has chronic diarrhea
* Has bowel dysfunction due to neurogenic disorder(s)
* Is in need of high-volume TAI (as estimated by investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Bowel function measured on a 10 cm Visual Analog Scale (VAS) at Baseline Visit (V1) and End of Clinical Investigation Visit (V7). | From enrollment to the end of treatment at week 12.
  0 cm = worst possible bowel function and 10 cm = best possible bowel function.

CONTACTS AND LOCATIONS:
Locations (1):
- Århus University Hospital, Aarhus, Gotland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided